CLINICAL TRIAL: NCT00451698
Title: Erythropoietin and Pediatric Cardiac Surgery
Acronym: EPO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate patient enrollment
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CHW 04/161
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Results first posted 2013-07-16 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Congenital Heart Defect
Keywords: Erythropoietin; Congenital heart surgery
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3 (Placebo Comparator): acyanotic placebo
  Interventions: Drug: acyanotic placebo
- 4 (Experimental): acyanotic erythropoietin
  Interventions: Drug: acyanotic erythropoietin

INTERVENTIONS:
Drug: acyanotic erythropoietin — Single dose IV push
  Arms: 4
Drug: acyanotic placebo — Single dose IV push
  Arms: 3

SUMMARY:
Lack of bloodflow to the heart and brain when the heart is stopped during heart surgery can cause damage to those organs. We hypothesize that a single dose of erythropoietin prior to the heart bypass portion of surgery may protect the infant human heart and brain from injury.

This randomized clinical trial will involve 120 children, age 6 weeks to 18 years, requiring heart bypass surgery for congenital heart defects.

DETAILED DESCRIPTION:
Lack of bloodflow to the heart and brain when the heart is stopped during heart surgery can cause damage to those organs. A medicine already used in humans, erythropoietin, may protect the heart and brain of children born with heart defects during their surgical repair. In a rabbit model, erythropoietin did protect the hearts. We hypothesize that a single dose of erythropoietin prior to the heart bypass portion of surgery may protect the infant human heart and brain from injury.

For this randomized control trial, 120 children, age 6 weeks to 18 years, requiring heart bypass surgery for congenital heart defects, will be divided into four groups. Two groups will be children whose usual blood oxygen level is low because of their heart defect; the other two will be children with normal blood oxygen levels. Each child will be randomized to receive either erythropoietin or placebo 15 minutes prior to stopping the heart during their surgery.

Erythropoietin's protective function will be measured after surgery by: (1) amount of medication required to support heart function, (2) how well the heart pumps blood as seen by echocardiogram, (3) levels of chemicals produced by the body when heart or brain tissue injury occurs, (4) urine output and oxygen levels (5) time on ventilator support (6) ICU stay and (7) hospital stay. Heart tissue will be collected during surgery to determine how erythropoietin protects heart cells.

Statistical tests including ANOVA will test for similarities and differences among the groups on the measures of protection from injury.

Note - the study design was edited after the FDA released a warning about the use of erythropoietin. Only acyanotic patients were recruited therefore only 2 study groups are included.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 weeks to 18 years
* Requiring open heart surgery for congenital heart defect -Parents able to speak English and document informed consent -

Exclusion Criteria:

* Received erythropoietin within past 30 days
* Previous adverse reaction to erythropoietin or to albumin
* History of neurological disorder -Laboratory evidence of kidney or liver dysfunction -

Ages: 6 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2007-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Zangwill, MD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin; John Baker, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Shi Y, Rafiee P, Su J, Pritchard KA Jr, Tweddell JS, Baker JE. Acute cardioprotective effects of erythropoietin in infant rabbits are mediated by activation of protein kinases and potassium channels. Basic Res Cardiol. 2004 May;99(3):173-82. doi: 10.1007/s00395-004-0455-x. Epub 2004 Jan 29. PMID 15088102

RESULTS

PARTICIPANT FLOW:
Groups:
- Acyanotic Placebo: Children requiring cardiac surgery with cardiopulmonary bypass with baseline saturations greater than 88% _ Received placebo
- Acyanotic Study Drug: Children requiring cardiac surgery with cardiopulmonary bypass with baseline saturations greater than 88% - Received study drug
Period: Overall Study
Arm/Group | Acyanotic Placebo | Acyanotic Study Drug
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acyanotic Placebo | Acyanotic Study Drug | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 6 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.1 (1.2) | 12.9 (4.5) | 9.6 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Markers of Heart Damage
Description: Troponin I levels (ng/ml) measured at 4 time points
Time Frame: 4 postoperative time points up to 48 hours
Population: Analysis was limited to descriptive statistics due to low enrollment and study closure.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Acyanotic Placebo | Acyanotic Study Drug
Number analyzed (Participants) | 3 | 6
ng/ml
  60 minutes post bypass | 31.1 (12.2) | 12.3 (9.2)
  4 hrs post bypass | 27.2 (8.6) | 15 (8.2)
  24 hrs post bypass | 10 (6.2) | 10.7 (10.4)
  48 hrs post bypass | 5.2 (1.9) | 5.2 (5.2)

2. Primary Outcome: Biochemical Markers of Neuron Damage
Time Frame: 4 postoperative time points
Population: There were 43 samples taken from the 9 subjects but no analysis was performed - the laboratory did not set up the assay to run the samples because the study did not have enough subjects to achieve statistical power.
Groups:
- Acyanotic Placebo: acyanotic placebo
  acyanotic placebo: Single dose IV push
- Acyanotic Erythropoietin: acyanotic erythropoietin
  acyanotic erythropoietin: Single dose IV push
Arm/Group | Acyanotic Placebo | Acyanotic Erythropoietin
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Echocardiographic Assessment of Heart Function
Time Frame: 24 hours postop
Population: These data were not collected.
Arm/Group | Acyanotic Placebo | Acyanotic Erythropoietin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Inotropic Support
Time Frame: 24 and 48 hours post operative
Population: These data were not collected
Arm/Group | Acyanotic Placebo | Acyanotic Erythropoietin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Length of Hospitalization
Time Frame: At hospital discharge, up to 30 days
Population: Analysis was limited to descriptive statistics due to low enrollment and study closure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Acyanotic Placebo | Acyanotic Study Drug
Number analyzed (Participants) | 3 | 6
days | 4.6 (1.2) | 6 (5.2)

ADVERSE EVENTS:
Arm/Group | Acyanotic Placebo | Acyanotic Study Drug
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 1/3 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyanotic Placebo (N=3) | Acyanotic Study Drug (N=6)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — A brief post -op seizure occurred in a study participant who received placebo. There were no clinical sequelae.

LIMITATIONS AND CAVEATS:
Analysis was limited to descriptive statistics due to low enrollment and study closure. The number of participants fell far short of study goals and the study was terminated prematurely due to inadequate enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes